CLINICAL TRIAL: NCT06259123
Title: Neoadjuvant [177Lu]Lu-PSMAI&T Radioligand Therapy (PSMA-RLT) for Patients With Oligometastatic Prostate Cancer Diagnosed Using [68Ga]Ga-PSMA-11 PET Imaging Followed by Radical Prostatectomy: A Prospective Phase II Pilot Study
Brief Title: Neoadjuvant PSMA-RLT in Oligometastatic PCa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sazan Rasul, MD, PhD, Physician and post-doctoral researcher, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1944/2022; 2022-004115-92 (EudraCT Number)
Record Dates: First submitted 2023-12-25; First posted 2024-02-14 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: [177Lu]Lu-PSMAI&T; Oligometastatic prostate cancer; Radical prostatectomy; Therapy toxicity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective single-center phase II study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oligometastatic prostate cancer diagnosed using [68Ga]Ga-PSMA-11 PET imaging (Experimental): Patients with oligometastatic PCa diagnosed using [68Ga]Ga-PSMA-11 imaging defined as M1a and/or M1b positive with ≤5 osseous metastases and/or M1c ≤3 lung metastases will receive 2 cycles of 5 GBq [177Lu]Lu-PSMA I&T at 6-week intervals prior radical prostatectomy.
  Interventions: Drug: [177Lu]Lu-PSMA I&T

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA I&T — 2 cycles of 5 GBq [177Lu]Lu-PSMA I&T at 6-week intervals prior radical prostatectomy for patients with oligometastatic prostate cancer
  Other Names: PSMA-RLT

SUMMARY:
Prospective single-center phase II study to evaluate the PSA, imaging and pathological response, as well as oncological outcomes of systemic radioligand therapy [177Lu]Lu-PSMAI&T (PSMA-RLT) in patients planned for radical prostatectomy (RP) for oligometastatic prostate cancer (PCa) diagnosed using [68Ga]Ga-PSMA-11 PET examination.

Ten patients with oligometastatic primary PCa diagnosed using [68Ga]Ga-PSMA-11 PET-CT/MRI imaging will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Oligometastatic PCa diagnosed using [68Ga]Ga-PSMA-11 imaging defined as M1a and/or M1b positive with ≤5 osseous metastases and/or M1c ≤3 lung metastases
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
* Patients must have adequate bone marrow reserve: WBC ≥1.5 x 109 /L, Platelets ≥100 x 109 /L and Haemoglobin ≥9 g/dL.
* Patients must have adequate renal function with eGFR ≥ 50mL/min/1.73m2 using the Modification of Diet Renal Disease (MDRD) equation and an Albumin level of ≥2.5 g/dL.
* Patients must be able to sign Informed Consent Form

Exclusion Criteria:

* Concomitant participation in any other interventional trial
* Concurrent severe oncologic and medical conditions that result in patients not having a life expectancy of longer than the duration of the trial.
* Nonmetastatic PCa on [68Ga]Ga-PSMA-11 imaging
* >5 osseous metastases on [68Ga]Ga-PSMA-11 imaging
* Visceral metastases, apart from lungs
* Age > 75 years.
* Ongoing or previous androgen deprivation therapy with agonist or antagonist therapies.
* Presence of clinically relevant somatic or psychiatric diseases that might interfere with the objectives and assessments of the study.
* Complete urinary out-flow obstruction or severe unmanageable urinary incontinence

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [Safety and Tolerability] of neoadjuvant PSMA-RLT and radical prostatectomy | 12 months
  Using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Furthermore, regular estimation of patient's ability to perform their usual everyday activities using Karnofsky performance status scale that ranges between a maximum of 100 percent (no restrictions) and 0 percent (death) and Eastern Cooperative Oncology Group Status scale that ranges from 0 (complete health) to 5 (death).

SECONDARY OUTCOMES:
PSA response to neoadjuvant PSMA-RLT and radical prostatectomy | 24 months
  in term of PSA decline of ≥ 50% from baseline value
Imaging response and stability to neoadjuvant PSMA-RLT and radical prostatectomy | 24 months
  in terms of disappearance of PSMA-avid lesions and/or size regression of the metastatic lymph nodes evaluated based on response evaluation criteria of solid tumor (RECIST) version 1.1.
Any therapy- and androgen deprivation therapy-free survival after radical prostatectomy, | 24 months
  estimate the time until the start of any therapy- and androgen deprivation therapy
Estimate time to castration-resistant prostate cancer | 24 months
  estimate the time until no PSA response in terms of PSA decline to androgen deprivation therapy
Evaluate pathologic response at radical prostatectomy | 24 months
  measured as rates of pathologic complete response, minimal residual disease, pT3 disease, positive surgical margins, and lymph node metastasis.
Quantification of circulating free tumor DNA (ctDNA) | 24 months
  enumeration of circulating tumor cells (CTCs) during the study period, molecular changes measured in liquid biopsy markers and tissue specimens following PSMA-RLT and radical prostatectomy and during follow-up.
Assess quality of life under the systemic PSMA-RLT | 24 months
  using the questionnaires: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) and Functional Assessment of Chronic Illness Therapy (FACT-P).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Upon request, we provide the individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For 2 years after the end of the trail